CLINICAL TRIAL: NCT05160402
Title: A Phase 1 Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Intranasal Plus Intraoral IGM-6268 in Healthy Volunteers
Brief Title: Evaluation of IGM-6268 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: IGM Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: IGM-6268-001
Record Dates: First submitted 2021-11-24; First posted 2021-12-16 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — IGM-6268

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive intranasal and intraoral administration of IGM-6268 or placebo at the assigned doses. Cohorts will be enrolled sequentially.
Who Masked: Participant, Investigator
Masking Description: Cohorts 1-6 will receive IGM-6268 or placebo. Subjects and Investigators will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (SAD) (Experimental): In Cohort 1, subjects will be randomized to receive a single intranasal and intraoral administration of 1 mg of IGM 6268 or placebo
  Interventions: Drug: IGM-6268; Drug: Placebo
- Cohort 2 (SAD) (Experimental): In Cohort 2, subjects will be randomized to receive a single intranasal and intraoral administration of 3.75 mg of IGM 6268 or placebo
  Interventions: Drug: IGM-6268; Drug: Placebo
- Cohort 3 (SAD) (Experimental): In Cohort 3, subjects will be randomized to receive a single intranasal and intraoral administration of 7.5 mg of IGM 6268 or placebo
  Interventions: Drug: IGM-6268; Drug: Placebo
- Cohort 4 (MAD) (Experimental): In Cohort 4, subjects will be randomized to receive a single intranasal and intraoral administration of 3.75 mg of IGM 6268 or placebo once a day for 5 days.
  Interventions: Drug: IGM-6268; Drug: Placebo
- Cohort 5 (MAD) (Experimental): In Cohort 5, subjects will be randomized to receive a single intranasal and intraoral administration of 7.5 mg of IGM 6268 or placebo once a day for 5 days.
  Interventions: Drug: IGM-6268; Drug: Placebo
- Cohort 6 (MAD) (Experimental): In Cohort 6, subjects will be randomized to receive a single intranasal and intraoral administration of 7.5 mg of IGM 6268 or placebo twice a day for 5 days.
  Interventions: Drug: IGM-6268; Drug: Placebo

INTERVENTIONS:
Drug: IGM-6268 — Active comparator
Drug: Placebo — Placebo comparator

SUMMARY:
This is a Phase 1, multi-center, randomized, double-blinded, placebo-controlled single (SAD) and multiple ascending (MAD) ascending dose study to assess the safety, tolerability, and pharmacokinetics (PK) of IGM-6268 administered intranasally and intraorally in healthy volunteers. IGM-6268 or placebo will be administered by intranasal + intraoral spray using a Teleflex Mucosal Atomization Device Nasal™ Intranasal Mucosal Atomization Device once (SAD), or once or twice each day for 5 days (MAD).

DETAILED DESCRIPTION:
IGM-6268 is an engineered Immunoglobulin M (IgM) antibody that specifically targets the receptor binding domain (RBD) of the SARS-CoV-2 spike protein. This humanized pentameric IgM antibody has 10 binding sites to the spike protein and a J-chain to enable the formation of IgM pentamers.

IGM-6268 is being developed as a treatment for or prophylaxis of symptoms associated with mild to moderate COVID-19. The primary mechanism of action of IGM-6268 is to block the binding of the SARS-CoV-2 RBD on the spike protein to human angiotensin converting enzyme 2 (hACE2), the cellular receptor for SARS-CoV-2. By blocking this binding, IGM 6268 neutralizes the infectivity of the virus.

ELIGIBILITY:
Inclusion Criteria:

* Is male or non-pregnant female adult ≥ 18 and ≤ 55 years of age
* Has a body mass index (BMI) < 35 kg/m2.
* Is healthy as determined by medical history, physical examination, 12-lead electrocardiogram, laboratory assessments, and vital signs at screening.
* For women of childbearing potential or men, agreement to use at least one highly effective form of non-hormonal contraception or one highly effective form and one effective form of non-hormonal contraception through the course of study treatment and for 3 months after the last dose of IGM-6268.
* Agrees to the collection of blood, urine, saliva, and nasopharyngeal samples, per protocol.

Exclusion Criteria:

* Receipt of any COVID-19 vaccine or contemplating receipt of any COVID-19 vaccine (or participating in a COVID-19 vaccine trial) during this study and follow-up periods (approximately 65 days from enrollment). Subjects are permitted to withdraw at any time if they decide to receive the vaccine
* History of prior positive SARS-CoV-2 diagnostic test (antigen or NAAT), or positive SARS-CoV-2 serology test, at any time before enrollment.
* Confirmed or suspected pulmonary or systemic bacterial infection.
* Current or planned participation in any interventional clinical trial during the study and follow-up periods.
* History of hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Uncontrolled human immunodeficiency virus (HIV) infection.
* Nasal polyps (history or physical exam) or any structural abnormality of nose that, in the opinion of the investigator, could compromise administration or receipt of study drug (e.g., nasal septal deviation).
* History of reactive airway disease or hypersensitivity to any component of study drug or placebo.
* Use of any nasally-administered drug between 5 days prior to study enrollment and 2 days after receipt of last dose administered.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability of IGM-6268 by assessing the number, severity, and type of adverse events per CTCAE 5.0 | Through 60 days following receipt of final dose

SECONDARY OUTCOMES:
IGM-6268 in serum | Predose through Day 3 (SAD) or Day 6 (MAD)
Incidence of anti-IGM-6268 antibodies in serum | Prior to dosing and at Day 28 following receipt of initial dose

CONTACTS AND LOCATIONS:
Overall Officials: Roel Funke, Study Director — IGM Biosciences, Inc.
Locations (1):
- Aventiv Research, Columbus, Ohio, United States